CLINICAL TRIAL: NCT06303661
Title: Non-ablative Radiofrequency and Low-intensity Shock Wave Therapy in Fibrotic Plaque in Men With Peyronie's Disease: Case Series
Brief Title: Non-ablative Radiofrequency and Low Intensity Shock Wave Therapy in Fibrotic Plaque in Men With Peyronie's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Atenção ao Assoalho Pélvico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 74001323.3.0000.5544
Record Dates: First submitted 2023-12-04; First posted 2024-03-12 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Peyronie Disease
Keywords: Peyronie Disease; Non ablative radiofrequency; Low-intensity Shock Waves Therapy
MeSH Terms: conditions — Penile Induration

STUDY DESIGN:
Intervention Model Description: Combination of two therapies with conservative devices is proposed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RF and SWT (Experimental): The treatment will be carried out through the application of monopolar non-ablative radiofrequency (IBRAMED, Amparo, São Paulo, Brazil - model Neartek) associated with electromagnetic low-intensity shock wave therapy (IBRAMED, Amparo, São Paulo, Brazil - model THOOR) on the fibrotic plaque in the penis, 2 to 5 times a week, according to the patient's availability, totaling 24 sessions.
  Interventions: Device: Non-ablative Radiofrequency; Device: Low-intensity Shock Wave Therapy

INTERVENTIONS:
Device: Non-ablative Radiofrequency — There are two electrodes: one active, which will be used on the penis, using a non-lubricated condom from the Blowtex brand, using pharmaceutical glycerin to emit radiofrequency inside and outside the condom, and another electrode, dispersive, wrapped in PVC-type plastic film, coupled to the region of the patient's penis where there is no fibrotic plaque, which will act as earth and the temperature to be used in the treatment will be 38°C. When the desired heating is reached, the device maintains the temperature and thus the radiofrequency application will be maintained for 2 minutes.
Device: Low-intensity Shock Wave Therapy — The equipment's applicator is covered with transparent PVC film and non-alcoholic gel is used as a coupling medium between the applicator and the penis. The following parameters are used: frequency of 10Hz, energy of 120mJ and 2,000 shots in the fibrotic plaque.

SUMMARY:
The goal of this one arm clinical trial is to evaluate the safety and describe the clinical response of non-ablative radiofrequency treatment associated with shockwave therapy in men with Peyronie's disease. The main question[s] it aims to answer are: • is the treatment safe? • is there any clinical response to the proposed treatment? Participants will respond to five validated questionnaires: International Index of Erectile Dysfunction (IIEF-5), Medical Outcomes Study 36 - Item Short - Form Health Survey (SF-36), Peyronie's Disease Questionnaire (PDQ), Scale Hospital for Anxiety and Depression (SHAD) and the Erection Quality Questionnaire (EQQ); will undergo a physical assessment that includes palpation of the fibrotic plaque on the penis, pharmacological induction of erection, and assessment of the size of the fibrotic plaque through ultrasound. Every five sessions, the participant's degree of satisfaction will be measured using a 5-point Likert scale, as well as the evolution of symptoms will also be observed, using a 10-point Visual Analogue Scale (VAS) and penile pain, if present. The entire evaluation protocol will be applied before (pre-test), after treatment (post-test) and 1 month after the end of treatment. Volunteers will be monitored by telephone to verify the long-term response after 3, 6, 9 and 12 months of completed treatment in relation to the Likert scale and VAS. The treatments they'll be given are • of monopolar non-ablative radiofrequency associated with • low-intensity shock wave therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical complaint related to Peyronie's disease;
* At any stage of the disease (acute or chronic).

Exclusion Criteria:

* Users of a pacemaker, cardiac defibrillator implant or any other electromagnetic implant;
* Metallic implants over or under the area to be treated.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
It is estimated that non-ablative RF associated with low-intensity SWT in patients with Peyronie Disease is a safe technique that leads to a satisfactory clinical response in relation to sexual function. | From enrollment to the end of treatment till 8 weeks, then at 1, 3, 6, 9 and 12 months.
  It will be measured by the questionnaire International Index of Erectile Dysfunction (IIEF-5). Lower values represent worse sexual function and are categorized as follows: 5-7 points represents severe erectile dysfunction, 8-11 points represents moderate erectile dysfunction, 12-16 represents mild to moderate erectile dysfunction, 17 -21 represents mild erectile dysfunction and 22-25 means no erectile dysfunction.
It is estimated that non-ablative RF associated with low-intensity SWT in patients with Peyronie Disease is a safe technique that leads to a satisfactory clinical response in relation to pain. | From enrollment to the end of treatment till 8 weeks, then at 1, 3, 6, 9 and 12 months.
  The level of pain will be assess by the question three questions of Peyronie's Disease Questionnaire (PDQ). Each of the three questions score from 0 to 10, so the total range will be from 0 to 30. The lower the score, the less pain the patient feels.
It is estimated that non-ablative RF associated with low-intensity SWT in patients with Peyronie Disease is a safe technique that leads to a satisfactory clinical response in relation to penile erection. | From enrollment to the end of treatment till 8 weeks, then at 1, 3, 6, 9 and 12 months.
  The quality of penile erection will be measured by the Quality of Erection Questionnaire. The final score can vary between 0 and 100 points, with the higher the score, the better the quality of the erection.

SECONDARY OUTCOMES:
It is estimated that non-ablative RF associated with low-intensity SWT in patients with Peyronie Disease is a technique that promotes a positive impact on quality of life and psycho-emotional aspects of anxiety and depression. | From enrollment to the end of treatment till 8 weeks, then at 1, 3, 6, 9 and 12 months.
  It will be measured by the questionnaire Medical Outcomes Study 36 - Item Short - Form Health Survey (SF-36). The final score for each domain ranges from 0 to 100 (there are two - body and mental), there is no cutoff point and higher scores indicate a better health status.
It is estimated that non-ablative RF associated with low-intensity SWT in patients with Peyronie Disease is a technique that promotes a positive impact on psycho-emotional aspects of anxiety and depression. | From enrollment to the end of treatment till 8 weeks, then at 1, 3, 6, 9 and 12 months.
  It will be measured by the questionnaire Scale Hospital for Anxiety and Depression. It is composed of two subscales, one for anxiety and the other for depression, with seven items each. The global score on each subscale ranges from 0 to 21. The lower the score, the lower level of anxiety/or depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Atenção ao Assoalho Pelvico, Salvador, Estado de Bahia, Brazil